CLINICAL TRIAL: NCT05542927
Title: Incidence of Acute Kidney Injury and Mortality in Critically Ill Patients: Urinary Chloride as a Prognostic Marker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdelrhman El shafei, M.B.B.CH., Ain Shams University
Other Study IDs: 541/2022
Record Dates: First submitted 2022-09-11; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill Acute kidney injury patients: AKI is defined as any of the following: Increase in SCr by ≥0.3 mg/dl (≥ 26.5 μmol/l) within 48 hours; OR increase in SCr to≥1.5 times baseline, which is known or presumed to have occurred within prior 7 days; OR Urine volume <0.5 ml/kg/h for 6 hour)
  1. Serum chloride, urinary chloride & serum creatinine will be requested on the first day of admission in ICU
  2. Serum chloride & urinary chloride will be requested every 48 hours in ICU with correlation between urinary chloride concentrations, AKI & mortality.
  3. Serum creatinine will be requested every 24 hours in ICU.
  4. Monitoring of Urinary Output every 24 hours.
  5. Daily SOFA score.
  Interventions: Diagnostic Test: urine chloride

INTERVENTIONS:
Diagnostic Test: urine chloride — Serum chloride, urinary chloride & serum creatinine will be requested on the first day of admission in Intensive Care Unit (ICU). 2. Serum chloride & urinary chloride will be requested every 48 hours in ICU with correlation between urinary chloride concentrations, AKI & mortality. 3. Serum creatinine will be requested every 24 hours in ICU. 4. Monitoring of Urinary Output (U.O.P.) every 24 hours

SUMMARY:
Acute kidney injury (AKI) is characterized by a rapid decrease in renal function. It is frequent in hospitalized patients and its incidence is higher in critically ill patients. It is associated with high rates of morbidity and mortality.

AKI affects over 13 million people per year globally, and results in 1.7 million deaths. It is diagnosed in up to 20% of hospitalized patients and in 30- 60% of critically ill patients. It is the most frequent cause of organ dysfunction in intensive care units and the occurrence of even mild AKI is associated with a 50% higher risk of death. AKI has been associated with longer hospital stays, in-hospital mortality, cardiovascular events, progression to chronic kidney disease and long-term mortality. It results in a significant burden for the society in terms of health resource use during the acute phase and the potential long-term sequelae including development of chronic kidney disease and kidney failure. Yunos et al. have focused on chloride, which is the most abundant strong anion in extracellular fluid. Progression of hyperchloremia in the ICU was identified as a predictor of increased mortality in a large retrospective cohort study of critically ill septic patients. Sadan et al. have shown associations between hyperchloremia and an increased incidence of AKI in patients with subarachnoid hemorrhage, as well as in patients who have undergone abdominal surgery. Abnormal blood chloride concentrations were associated with metabolic acidosis, which may worsen patient outcomes. Moreover, hyperchloremia may be caused by inappropriate fluid management with chloride-rich solutions.

Importantly, chloride-rich solutions were reportedly associated with hyperchloremia and major adverse kidney disease, including death, in intensive care settings. Urine samples are relatively easy to collect in ICU, and real-time urinary electrolyte monitoring device is available for clinical use. In addition, recent development of urinary AKI biomarkers has enabled clinical evaluation of kidney function. Komaru et al. examined associations among urinary chloride, mortality, and AKI incidence in ICU patients and concluded that lower urinary chloride concentration was associated with increased mortality and incidence of AKI in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 years old and above.
* No history of chronic kidney disease (CKD).

Exclusion Criteria:

* Age under 21 years old.
* Patients leaving the ICU within 24 hours for any reason.
* Anuric patients.
* Patients on maintenance hemodialysis.
* Patients those without day 1 urinary or blood tests.
* Refusal of patient or his/her relative participation in the study

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients diagnosed with AKI
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuarcy of urinary chloride for incidence of AKI | 10 days
  correlation between urinary chloride concentrations and incidence of AKI.

SECONDARY OUTCOMES:
28-day mortality | 28 days
  correlation between urinary chloride concentrations and mortality of AKI patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Ain shams university., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: contact principal investigators

REFERENCES:
- [Background] Kellum JA, Prowle JR. Paradigms of acute kidney injury in the intensive care setting. Nat Rev Nephrol. 2018 Apr;14(4):217-230. doi: 10.1038/nrneph.2017.184. Epub 2018 Jan 22. PMID 29355173
- [Background] Abd ElHafeez S, Tripepi G, Quinn R, Naga Y, Abdelmonem S, AbdelHady M, Liu P, James M, Zoccali C, Ravani P. Risk, Predictors, and Outcomes of Acute Kidney Injury in Patients Admitted to Intensive Care Units in Egypt. Sci Rep. 2017 Dec 7;7(1):17163. doi: 10.1038/s41598-017-17264-7. PMID 29215080
- [Background] Hoste EAJ, Kellum JA, Selby NM, Zarbock A, Palevsky PM, Bagshaw SM, Goldstein SL, Cerda J, Chawla LS. Global epidemiology and outcomes of acute kidney injury. Nat Rev Nephrol. 2018 Oct;14(10):607-625. doi: 10.1038/s41581-018-0052-0. PMID 30135570
- [Background] Yunos NM, Bellomo R, Story D, Kellum J. Bench-to-bedside review: Chloride in critical illness. Crit Care. 2010;14(4):226. doi: 10.1186/cc9052. Epub 2010 Jul 8. PMID 20663180
- [Background] Neyra JA, Canepa-Escaro F, Li X, Manllo J, Adams-Huet B, Yee J, Yessayan L; Acute Kidney Injury in Critical Illness Study Group. Association of Hyperchloremia With Hospital Mortality in Critically Ill Septic Patients. Crit Care Med. 2015 Sep;43(9):1938-44. doi: 10.1097/CCM.0000000000001161. PMID 26154934
- [Background] Sadan O, Singbartl K, Kandiah PA, Martin KS, Samuels OB. Hyperchloremia Is Associated With Acute Kidney Injury in Patients With Subarachnoid Hemorrhage. Crit Care Med. 2017 Aug;45(8):1382-1388. doi: 10.1097/CCM.0000000000002497. PMID 28504980
- [Background] Semler MW, Self WH, Wanderer JP, Ehrenfeld JM, Wang L, Byrne DW, Stollings JL, Kumar AB, Hughes CG, Hernandez A, Guillamondegui OD, May AK, Weavind L, Casey JD, Siew ED, Shaw AD, Bernard GR, Rice TW; SMART Investigators and the Pragmatic Critical Care Research Group. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):829-839. doi: 10.1056/NEJMoa1711584. Epub 2018 Feb 27. PMID 29485925